CLINICAL TRIAL: NCT02611076
Title: Expanding the Reach of a Validated Smoking-Cessation Intervention: A Spanish-Language Clinical Trial
Brief Title: Smoking-cessation: A Spanish-Language Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: James and Esther King Biomedical Research Program (Other); University of Miami (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: MCC-18231
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Smoking Cessation; Tobacco Dependence
Keywords: smoking cessation; self-help; Spanish language
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stop Smoking for Good Intervention in Spanish (Experimental): Study II: Stop Smoking for Good Intervention in Spanish (SS-SP) will comprise a series of 10 booklets distributed over 18 months, plus additional monthly contacts via 9 supportive pamphlets developed in Study I. Behavioral: Stop Smoking for Good Intervention in Spanish (SS-SP) Assessments will occur at six-month intervals, through 24 months.
  Interventions: Behavioral: Stop Smoking for Good Intervention in Spanish (SS-SP)
- Usual Care (Active Comparator): Study II: Usual Care (UC) will comprise a single, Spanish-language, smoking cessation booklet developed by the National Cancer Institute (NCI). Behavioral: Usual care (UC) Assessments will occur at six-month intervals, through 24 months.
  Interventions: Behavioral: Usual care (UC)

INTERVENTIONS:
Behavioral: Stop Smoking for Good Intervention in Spanish (SS-SP) — Assessments will occur at six-month intervals, through 24 months.
  Arms: Stop Smoking for Good Intervention in Spanish
Behavioral: Usual care (UC) — Assessments will occur at six-month intervals, through 24 months.
  Arms: Usual Care

SUMMARY:
The purpose of this study is to develop and test a series of culturally relevant and appropriate booklets in Spanish, designed to assist Hispanic smokers in quitting smoking and remaining smoke-free.

DETAILED DESCRIPTION:
Study Aim 1: To transcreate the existing English-language 10 "Stop Smoking for Good" booklets and accompanying 9 supportive "My Story" pamphlets into a series of culturally relevant and acceptable materials for Spanish-speaking smokers who prefer to receive health information in Spanish. The adaptation of the intervention materials will be based upon the findings from a systematic formative evaluation employing a heterogeneous group of Hispanic/Latino smokers representing diverse subcultural groups.

Study Aim 2: To test the efficacy of the self-help intervention developed in Study I among Spanish-speaking smokers in a randomized controlled trial. Participants (500) will be randomized to receive the Spanish-language version of the Stop Smoking for Good (SS-SP) intervention or usual care (UC) comprising an existing booklet from NCI. Investigators hypothesize SS-SP will produce higher abstinence rates than UC through 24 months.

Secondary Aim: Test moderator variables to improve targeting the intervention. Moderator analyses will be exploratory, without strong a priori hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* All Except Study I; Phase I Focus Group: monolingual Spanish, or bilingual Spanish-English and prefer receiving educational health materials in Spanish.
* Study I; Phase I Focus Group Only: Able to speak and read in English and Spanish.
* ≥ 1 year history of smoking
* Smoking ≥ 5 cigarettes per week
* Age ≥ 18 years
* Not currently enrolled in a face-to-face smoking cessation program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2016-10-11 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Study I: Completion of the Development of the Spanish Language Version of Smoking Cessation Materials | Up to 12 months
  Complete formative research, including focus groups and learner verification interviews to adapt Spanish language intervention materials in preparation for a randomized controlled trial.
Study II: Rate of Smoking Cessation | Up to 24 months
  Smoking cessation rates based on 7-day-point-prevalence abstinence (not smoking at all for 7 consecutive days) per study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Vani N. Simmons, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/